CLINICAL TRIAL: NCT02140788
Title: A Comparison Of The Effects Of Added Metformin (Versus No Added Metformin) On Psychopathology, Lipids, And Measures of Inflammation During The Initiation Or Re-Institution Of Treatment With Clozapine In Patients With Schizophrenia Or Schizoaffective Disorder
Brief Title: Effects of Metformin and Fish Oil on Treatment With Clozapine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: Pro00027822
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2014-05

CONDITIONS: Schizophrenia; Schizo-affective Disorder
Keywords: schizophrenia; schizo-affective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Metformin; Fish Oils

ARMS (4):
- Metformin (Active Comparator): Subjects will continue to take the clozapine prescribed as standard of care. Subjects assigned to added metformin will receive metformin 250 mg BID days 1-3, 500 mg BID days 4-7, and 1000 mg BID days 8-28 with breakfast and supper. Patients unable to tolerate a dose escalation will have the metformin dose reduced to the previously tolerated lower dose.
  Interventions: Drug: Metformin
- Fish Oil (Active Comparator): Subjects will continue to take the clozapine prescribed as standard of care. Subjects assigned to added fish oil will receive OmegaBrite 500 mg gel cap BID days 1-7, and 1000 mg BID days 8-28 with breakfast and supper. Patients unable to tolerate the dose escalation to 1000 mg BID will have the fish oil dose reduce to 500 mg BID.
  Interventions: Drug: Fish Oil
- Metformin and Fish Oil (Active Comparator): Subjects will continue to take the clozapine prescribed as standard of care. Subjects will receive Metformin and Fish Oil as part of the study.
  Interventions: Drug: Metformin; Drug: Fish Oil
- No medication added (No Intervention): Subjects will continue to take the clozapine prescribed as standard of care. Subjects will not receive Metformin or Fish Oil.

INTERVENTIONS:
Drug: Metformin
  Arms: Metformin; Metformin and Fish Oil
Drug: Fish Oil
  Arms: Fish Oil; Metformin and Fish Oil

SUMMARY:
One purpose of this study is to test whether adding metformin will limit some of the unwanted effects of clozapine, compared to not adding metformin. Metformin is a medication that is approved by the United States Food and Drug Administration (FDA) for the treatment of type-2 diabetes. Studies have found that people with type-2 diabetes often lose some weight when they take metformin, however the FDA has not approved metformin for weight loss, so for this study the use of metformin is investigational. This study will test whether metformin can help people with schizophrenia or schizoaffective disorders lose weight.

Another purpose of this study is to test whether adding fish oil will improve the benefit of clozapine and/or limit some of the unwanted effects of clozapine, compared to not adding fish oil. Fish oil is a medication used to reduce levels of some fats (triglycerides) in blood. Some studies have found that adding fish oil reduces psychosis (voices, suspiciousness). However the FDA has not approved fish oil for reducing psychosis, so for this study the use of fish oil is investigational. This study will test whether fish oil can help people with schizophrenia or schizoaffective disorders have less psychosis. Fish oil is not an antipsychotic medication.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients with clinical diagnoses of schizophrenia or schizo-affective disorder
* between 18 and 60 years of age
* patients whose treating clinicians have recommended treatment with clozapine (and the patients have agreed and provided signed informed consent for treatment with clozapine)

Exclusion Criteria:

* patients who have contraindications to metformin use, such as:

  * a diagnosis of congestive heart failure
  * renal impairment (serum creatinine > 1.5 in males; > 1.4 in females)
  * hepatic disease (AST or ALT > 2.0 times upper limit of normal (ULN)
  * positive hepatitis B surface antigen or hepatitis C antibody
  * total bilirubin>1.2x ULN; majority conjugated
  * metabolic acidosis (serum CO2 < lower limit of normal),
  * known hypersensitivity to metformin,
  * recent (in the past 30 days) or scheduled radiological studies involving iodinated contrast material
  * alcohol abuse/dependence within the past month
  * concurrent treatment with drugs that are known to increase metformin blood levels including furosemide, nifedipine, and cationic drugs including cimetidine, amiloride, digoxin, morphine, procainamide, quinidine, ranitidine, triamterene, trimethoprim, and vancomycin
* patients with blood dyscrasias that could be worsened by added fish oil
* women who are pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McEvoy, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-four subjects were consented to the study; however, were never randomized. The study was terminated in Feb 2013 and no data was collected or analyzed.
Groups:
- Metformin: Subjects will continue to take the clozapine prescribed as standard of care. Subjects assigned to added metformin will receive metformin 250 mg BID days 1-3, 500 mg BID days 4-7, and 1000 mg BID days 8-28 with breakfast and supper. Patients unable to tolerate a dose escalation will have the metformin dose reduced to the previously tolerated lower dose.
  Metformin
- Fish Oil: Subjects will continue to take the clozapine prescribed as standard of care. Subjects assigned to added fish oil will receive OmegaBrite 500 mg gel cap BID days 1-7, and 1000 mg BID days 8-28 with breakfast and supper. Patients unable to tolerate the dose escalation to 1000 mg BID will have the fish oil dose reduce to 500 mg BID.
  Fish Oil
- Metformin and Fish Oil: Subjects will continue to take the clozapine prescribed as standard of care. Subjects will receive Metformin and Fish Oil as part of the study.
  Metformin
  Fish Oil
Period: Overall Study
Arm/Group | Metformin | Fish Oil | Metformin and Fish Oil | No Medication Added
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who signed a consent form
Groups:
- All Subjects Who Consented: All subjects who signed a consent form
Arm/Group | All Subjects Who Consented
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Time Frame: baseline, 2 weeks, 4 weeks
Population: Patients were not randomized per protocol and the study was terminated. Data analysis was not performed.
Arm/Group | Metformin | Fish Oil | Metformin and Fish Oil | No Medication Added
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Changes in Fasting Levels of Non-HDL Cholesterol and Triglycerides
Time Frame: baseline, 2 weeks, 4 weeks
Population: Patients were not randomized per protocol and the study was terminated. Data analysis was not performed.
Arm/Group | Metformin | Fish Oil | Metformin and Fish Oil | No Medication Added
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Changes in C-reactive Protein and Sedimentation Rates
Time Frame: baseline, 2 weeks, 4 weeks
Population: Patients were not randomized per protocol and the study was terminated. Data analysis was not performed.
Arm/Group | Metformin | Fish Oil | Metformin and Fish Oil | No Medication Added
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Changes in Mole Percentages of Omega-3 PUFAs in Fasting Serum and RBC Membranes
Time Frame: baseline, 2 weeks, 4 weeks
Population: Patients were not randomized per protocol and the study was terminated. Data analysis was not performed.
Arm/Group | Metformin | Fish Oil | Metformin and Fish Oil | No Medication Added
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Changes in Total Scores on the 4 Positive Brief Psychiatric Rating Scale (BPRS) Items
Description: The four positive items are: Suspiciousness, Unusual Thought Content, Hallucinations, Conceptual Disorganization.
Time Frame: baseline, 2 weeks, 4 weeks
Population: Patients were not randomized per protocol and the study was terminated. Data analysis was not performed.
Arm/Group | Metformin | Fish Oil | Metformin and Fish Oil | No Medication Added
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Metformin | Fish Oil | Metformin and Fish Oil | No Medication Added
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Patients were not randomized per protocol and the study was terminated. Data analysis was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes